CLINICAL TRIAL: NCT05417763
Title: Pressure Microcatheter for Physiological Measurements - A Prospective, Multicenter, Randomized Study
Brief Title: Sensor-equipped Ultrathin Pressure Microcatheter Versus Pressure Wire for Physiological Measurements
Acronym: SUPREME II
Status: Completed | Type: Observational
Sponsor: Insight Lifetech Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other); Peking University Third Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Sir Run Run Shaw Hospital (Other); Shandong Provincial Hospital (Other Government); Zunyi Medical College (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CTP-01-001
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia
Keywords: fractional flow reserve; constant-resistance ratio; resting full-cycle ratio
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pressure Microcatheter-First: Per the result of prior randomization, physiological assessment to the enrolled patient will be performed by the TruePhysio pressure microcatheter system ahead of the Pressure Wire system.
  Interventions: Device: Randomized physiological measurements by the two systems
- Pressure Wire-First: Per the result of prior randomization, physiological assessment to the enrolled patient will be performed by the Pressure Wire system ahead of the TruePhysio pressure microcatheter system, per the result of prior randomization.
  Interventions: Device: Randomized physiological measurements by the two systems

INTERVENTIONS:
Device: Randomized physiological measurements by the two systems — To measure physiological indices (FFR, cRR and RFR), either pressure microcatheter or pressure wire enters one patient's body. Whether it is the pressure microcatheter or pressure wire firstly to enter is randomized. After completion of one system's physiological assessment, the other system will follow for its physiological assessment.

SUMMARY:
TruePhysio pressure microcatheter is a novel device for evaluating the functional significance of coronary stenosis, and its safety and efficacy on the measurement of hyperemic index have been validated in the previous SUPREME study (NCT03541577). This study will further evaluate the safety and efficacy of the physiological indices measured by the TruePhysio pressure microcatheter, including resting and hyperemic indices, with respect to the physiological indices measured by the Pressure Wire.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of the constant-resistance ratio (cRR) measured by the TruePhysio pressure microcatheter, in both binary and hybrid strategy, with respect to its own fractional flow reserve (FFR) and the FFR or resting full-cycle ratio (RFR) by the Pressure Wire. And the safety and efficacy of the FFR measured by the TruePhysio pressure microcatheter in patients with a border range of diameter stenosis also be validated with respect to the FFR by the Pressure Wire.

The diagnostic accuracy of cRR by the TruePhysio pressure microcatheter system is evaluated, using FFR measured by both systems as reference;

Mean bias between the FFR values measured by TruePhysio pressure microcatheter and Pressure Wire is evaluated, using FFR measured by Pressure Wire as the reference;

The diagnostic accuracy of the hybrid cRR-FFR scheme by the TruePhysio pressure microcatheter is evaluated, using its own FFR as reference;

The diagnostic accuracy of the hybrid RFR-FFR scheme by the Pressure Wire system is evaluated, using its own FFR as reference.

The hybrid scheme for cRR-FFR (pressure microcatheter system), or RFR-FFR (pressure wire system), is defined as following:

* the gray zone is defined as where the sensitivity and specificity are equal, shown as [A, B].
* if cRR or RFR of the target vessel is <A, it is diagnosed as functionally positive in myocardial ischemia;
* if cRR or RFR of the target vessel is >B, it is diagnosed as functionally negative in myocardial ischemia;
* if cRR or RFR of the target vessel is between A and B (including A and B), the diagnostic criterion is superseded by that of FFR, which is:

  * if FFR of the target vessel is > 0.80, it is diagnosed as functionally negative in myocardial ischemia;
  * if FFR of the target vessel is ≤ 0.80, it is diagnosed as functionally positive in myocardial ischemia.

A total of 487 patients are anticipated to be recruited from 11 centers in China.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Having at least one 30-90% coronary artery stenosis by visual estimation under angiogram;
* Clinically indicated to physiological assessment.

Exclusion Criteria:

* Unable to comprehend, or unwilling to sign the informed consent form;
* Contraindicated to the procedures of invasive coronary angiography or percutaneous coronary intervention;
* Clinically diagnosed with severe coronary artery vasospasm;
* Other operator-discerned facts that will make enrollment or the procedure impossible to complete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of cRR measured by TruePhysio pressure microcatheter in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by TruePhysio pressure microcatheter as the reference. The optimal binary cutoff for cRR is determined by using Youden's index.

SECONDARY OUTCOMES:
The area under the Receiver Operating Characteristic (ROC) curve (AUC) of cRR measured by the TruePhysio pressure microcatheter in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by TruePhysio pressure microcatheter as the reference
The sensitivity, specificity, positive and negative predictive values of cRR measured by TruePhysio pressure microcatheter in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by TruePhysio pressure microcatheter as the reference. The optimal binary cutoff for cRR is determined by using Youden's index.
The AUC of cRR measured by the TruePhysio pressure microcatheter in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference
The overall accuracy, sensitivity, specificity, positive and negative predictive values of cRR in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference. The optimal binary cutoff for cRR is determined by using Youden's index.
The AUC of RFR measured by the Pressure Wire in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference
The overall accuracy, sensitivity, specificity, positive predictive value and negative predictive value of RFR in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference. The binary cutoff for RFR is determined by previous study as 0.89.
The overall accuracy, sensitivity, specificity, positive and negative predictive values of the hybrid cRR-FFR scheme, concluded by TruePhysio pressure microcatheter, in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the TruePhysio pressure microcatheter as the reference. The gray zone is defined as where the false positive and negative ratios are equal.
The proportion of the subcohort, whose cRR value is in the gray zone of the hybrid cRR-FFR scheme, to the entire cohort | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the TruePhysio pressure microcatheter as the reference. Each enrolled patient only has one vessel to be physiologically assessed.
When the cRR value is out of the gray zone of the hybrid cRR-FFR scheme, the cRR-FFR hybrid scheme's accuracy in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the TruePhysio pressure microcatheter as the reference
The overall accuracy, sensitivity, specificity, positive and negative predictive values of the hybrid RFR-FFR scheme, concluded by Pressure Wire, in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the Pressure Wire as the reference. The gray zone is determined by previous study as [0.86, 0.93].
The proportion of the subcohort, whose RFR value is in the gray zone of the hybrid RFR-FFR scheme, to the entire cohort | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the Pressure Wire as the reference. Each enrolled patient only has one vessel to be physiologically assessed.
When the RFR value is out of the gray zone of the hybrid RFR-FFR scheme, the RFR-FFR hybrid scheme's accuracy in diagnosing myocardial ischemia | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by the Pressure Wire as the reference
Results of Pearson correlation between the cRR and FFR measured by TruePhysio pressure microcatheter | Immediate upon completion of the procedure for the last enrolled patient
  Paired values are analyzed by Pearson correlation
Results of Passing-Bablok regression analysis between the cRR and FFR measured by TruePhysio pressure microcatheter | Immediate upon completion of the procedure for the last enrolled patient
  Paired values are analyzed by Passing-Bablok regression
Results of Pearson correlation between the RFR and FFR measured by Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired values are analyzed by Pearson correlation
Results of Passing-Bablok regression analysis between RFR and FFR measured by Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired values are analyzed by Passing-Bablok regression
Results of Passing-Bablok regression analysis between cRR measured by the TruePhysio pressure microcatheter, and RFR measured by the Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired cRR-RFR values by the two systems are analyzed in Passing-Bablok regression
Results of Bland-Altman analysis between cRR measured by the TruePhysio pressure microcatheter, and RFR measured by the Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired cRR-RFR values by the two systems are analyzed in Bland-Altman analysis
Results of Pearson's correlation between cRR measured by the TruePhysio pressure microcatheter, and RFR measured by the Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired cRR-RFR values by the two systems are analyzed in Pearson correlation
Results of Pearson correlation between the FFR values measured by TruePhysio pressure microcatheter and Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired FFR values by the two systems are analyzed by Pearson correlation
Results of Passing-Bablok regression analysis between the FFR values measured by TruePhysio pressure microcatheter and Pressure Wire | Immediate upon completion of the procedure for the last enrolled patient
  Paired FFR values by the two systems are analyzed by Passing-Bablok regression
Mean bias between the FFR values measured by TruePhysio pressure microcatheter and Pressure Wire as assessed by Bland-Altman analysis | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference
Results of Bland-Altman analysis between the FFR values measured by TruePhysio pressure microcatheter and Pressure Wire among the patients with atrial fibrillation or in severe stenosis or with small vessels | Immediate upon completion of the procedure for the last enrolled patient
  Using FFR measured by Pressure Wire as the reference. The severe stenosis is defined as the diameter stenosis higher than 70%, while the small vessel is defined as the reference vessel diameter smaller than 2.5 mm.
Rate of significant drift | Immediate upon completion of the procedure for the last enrolled patient
  Drift is defined as the difference between FFR value and 1 when pressure sensor is pulled back to coronary artery ostium for verification.
  Significant drift occurs when the device has a drift with absolute value > 0.03; alternatively, drift is regarded as significant when the Pd/Pa at the ostium for verification is either <0.97 or >1.03.
  Significant drift is recorded per appearance, regardless whether the measurement is eventually successful or not. Its rate is calculated as:
  Times of significant drift occurred in total / Times of measuring attempted in total
Rate of device success | Immediate upon completion of the procedure for the last enrolled patient
  Device success is defined when a device successfully crossed the lesion and completed acquisition of valid physiological values.
  For any vessel, if valid cRR and FFR values by the TruePhysio pressure microcatheter are acquired, the measurement of TruePhysio pressure microcatheter is successful in the specific vessel, disregarding how many times it was attempted;
  For any vessel, if valid RFR and FFR values by the Pressure Wire are acquired, the measurement of Pressure Wire is successful in the specific vessel, disregarding how many times it was attempted.
  Rate of device success is calculated as:
  Vessels with device success / Total vessels

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang